CLINICAL TRIAL: NCT05740332
Title: Wet Time for a Foam Hand Sanitizer With 70% Ethyl Alcohol
Brief Title: Wet Time for a Foam Hand Sanitizer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medline Industries (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MED-2022-DIV60-002
Record Dates: First submitted 2023-02-13; First posted 2023-02-23 (Actual); Results first posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Hand Hygiene Effectiveness
MeSH Terms: interventions — Ethanol

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- All participants (Experimental): 1 mL of alcohol foam hand sanitizer automatically dispensed into hands, spread over hands and rubbed until dry.
  Interventions: Drug: Alcohol hand sanitizer foam

INTERVENTIONS:
Drug: Alcohol hand sanitizer foam — 1mL of alcohol foam hand sanitizer automatically dispensed into hands, spread over hands and rubbed until dry.
  Other Name: Medline Spectrum™ Advanced Hand Sanitizer Foam (70%)

SUMMARY:
Hand sanitizers are a standard of hygiene requirements. They must be effective at reducing germ count on the hands while ideally providing emollients to moisturize the skin after use. Spectrum™ Advanced Hand Sanitizer Foam (70%) (hereby referred to as Spectrum Advanced Foam) kills over 99.99% of germs within 15 seconds while boasting double digit increases in hand moisture after two weeks of use.

In 2002 and 2009 the Center for Disease Control and Prevention (CDC) and World Health Organization (WHO) published guidance that hands should remain wet for at least 15 seconds while being rubbed together after application of an alcohol-based hand rub, though the recommendations do not specify the volume of product to be apply.

This study will evaluate the "wet time" of Spectrum Advanced Foam, which will be defined as the length of time in which the sanitizer foam stays wet on the hands while the participant rubs their hands with the foam sanitizer. The participant will first be asked to wash and dry their hands. Participants will review the appropriate hand sanitizer application steps, as detailed by the WHO guidance. Then, a 1.0 milliliter (mL) aliquot of Spectrum Advanced Foam will be dispensed from an automated dispenser to the participant's hands. The participant will be asked to rub their hands together following the WHO method for hand sanitizer application until they declare the product has dried sufficiently for the donning of medical gloves. Study personnel will measure the wet time of Spectrum Advanced foam using a stopwatch. If the 1.0 ml aliquot does not yield sufficient results to meet WHO guidelines then a 1.4 ml aliquot will be tested, however this was not the case for our study.

DETAILED DESCRIPTION:
Hand sanitizers are a standard of hygiene requirements. They must be effective at reducing germ count on the hands while ideally providing emollients to moisturize the skin after use. In 2002 and 2009 the CDC and WHO published guidances that hands should remain wet for at least 15 seconds while being rubbed together after application of an alcohol-based hand rub, though the recommendations do not specify the volume of product to be apply. The CDC specifically recommends applying alcohol-based hand sanitizers by applying the manufacturer-recommended amount of sanitizer directly to the palm of one hand and then rubbing the hands together. The sanitizer must entirely cover the surfaces of both hands and all fingers while rubbing the hands together until the product has dried. The goal of this study is to evaluate the "wet time" of Spectrum Advanced Foam, which will be defined in this study as the length of time in which the foam sanitizer stays wet on the hands while the participant rubs their hands with the foam sanitizer.

ELIGIBILITY:
Inclusion Criteria:

* Individual ≥ 18 years of age

Exclusion Criteria:

* Individual has a self reported skin condition that might result in irritation from the hand sanitizer.
* Individual has a known allergy to the ingredients in the test product.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2023-01-12 (Actual); Study Completion 2023-01-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medline Industries, LP, Northfield, Illinois, United States

REFERENCES:
- [Result] Boyce JM, Pittet D; Healthcare Infection Control Practices Advisory Committee; HICPAC/SHEA/APIC/IDSA Hand Hygiene Task Force. Guideline for Hand Hygiene in Health-Care Settings. Recommendations of the Healthcare Infection Control Practices Advisory Committee and the HICPAC/SHEA/APIC/IDSA Hand Hygiene Task Force. Society for Healthcare Epidemiology of America/Association for Professionals in Infection Control/Infectious Diseases Society of America. MMWR Recomm Rep. 2002 Oct 25;51(RR-16):1-45, quiz CE1-4. PMID 12418624
- [Result] WHO Guidelines on Hand Hygiene in Health Care: First Global Patient Safety Challenge Clean Care Is Safer Care. Geneva: World Health Organization; 2009. Available from http://www.ncbi.nlm.nih.gov/books/NBK144013/ PMID 23805438

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: 1 mL of alcohol foam hand sanitizer automatically dispensed into hands, spread over hands and rubbed until dry.
  Alcohol hand sanitizer foam: 1mL of alcohol foam hand sanitizer automatically dispensed into hands, spread over hands and rubbed until dry.
  Other Name: Medline Spectrum™ Advanced Hand Sanitizer Foam (70%)
Period: Overall Study
Arm/Group | All Participants
Started | 46
Completed | 46
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 46
Age, Continuous [Mean (Full Range); unit: years] | 34.6 [23 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Foam Sanitizer Wet Time Duration
Description: To determine the duration of time during which a 1.0 mL aliquot of Spectrum Advanced Hand Sanitizer Foam remains wet under conventional use conditions.
Time Frame: 2 mins
Population: 46 healthy adult participants
Measure: Mean (Standard Deviation); unit: time in seconds
Arm/Group | All Participants
Number analyzed (Participants) | 46
time in seconds | 35.41 (13.51)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/46
Serious Adverse Events (participants affected / at risk) | 0/46
Other Adverse Events (participants affected / at risk) | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-18): https://cdn.clinicaltrials.gov/large-docs/32/NCT05740332/Prot_SAP_000.pdf